CLINICAL TRIAL: NCT06264739
Title: Comparison of the Effects of Remifentanil and Dexmedetomidine on Postoperative Acute Pain in Patients Who Received Erector Spina Plane Block in Spinal Surgeries
Brief Title: Erector Spinae Block -Dexmedetomidine
Acronym: esp -dex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, ferdi gülaştı, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 22-12-23/2
Record Dates: First submitted 2023-12-22; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Acute Pain; Opioid Consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Remifentanil

STUDY DESIGN:
Intervention Model Description: randomized double blinding
Who Masked: Participant, Care Provider
Masking Description: Blindness patients and those who follow up after surgery will not know which group is in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Other): Dexmedetomidine (dekstomid) infusion will be administered for intraoperative analgesia.
  Interventions: Drug: esp Dexmedetomidine (dekstomid)
- group 2 (Other): remifentanyl (ultiva) infusion will be administered for intraoperative analgesia.
  Interventions: Drug: esp remifentanyl (ultiva)

INTERVENTIONS:
Drug: esp Dexmedetomidine (dekstomid) — After anesthesia and surgical procedures, bilateral ESP block will be applied under ultrasonography guidance from the midline 3 cm lateral from the T10 level. After cleaning the area with povidone-iodine before the block, the T10 transverse protrusion will be determined using a linear ultrasound probe. Local anesthetic will be applied between the transverse process and the erector spinae muscle with the help of an insulated needle designed for peripheral block procedures. The location of the needle will be confirmed by hydrodissection with physiological saline without local anesthesia. After the location of the needle is confirmed, 20 ml of LA and saline mixture will be applied and the same process will be repeated in the contralateral side. Of the total 40 ml LA, 20 ml will consist of bupivacaine 0.5% (marcaine), 10 ml will consist of lidocaine 2% (aritmal), and 10 ml will consist of physiological saline.
  Arms: group 1
Drug: esp remifentanyl (ultiva) — After anesthesia and surgical procedures, bilateral ESP block will be applied under ultrasonography guidance from the midline 3 cm lateral from the T10 level. After cleaning the area with povidone-iodine before the block, the T10 transverse protrusion will be determined using a linear ultrasound probe. Local anesthetic will be applied between the transverse process and the erector spinae muscle with the help of an insulated needle designed for peripheral block procedures. The location of the needle will be confirmed by hydrodissection with physiological saline without local anesthesia. After the location of the needle is confirmed, 20 ml of LA and saline mixture will be applied and the same process will be repeated in the contralateral side. Of the total 40 ml LA, 20 ml will consist of bupivacaine 0.5% (marcaine), 10 ml will consist of lidocaine 2% (aritmal), and 10 ml will consist of physiological saline.
  Arms: group 2

SUMMARY:
Postoperative pain is common after spinal surgeries, including lumbar disc surgery. Surgical anesthesia and perioperative analgesic regimen are aimed at complete intraoperative amnesia, deep analgesia, effective control of autonomic responses and rapid discharge from the hospital.

Although there are many studies on the use of these techniques for postoperative analgesia, the number of data comparing these techniques that can be used in meta-analyses is low. In our study, investigators aimed to compare the effects of remifentanil and dexmedetomidine accompanied by ESP block, which are different multimodal analgesia methods, on pain.

DETAILED DESCRIPTION:
investigators propose a randomized double-blind study comparing the use of intraoperative dexmedetomidine (Group D) for analgesic purposes with the use of intraoperative remifentanil (Group R) in patients undergoing ESP block for spinal surgery.

The clinic's routine anesthesia protocol will be applied to the patient. Anesthesia will not be interfered with.

Group 1: Dexmedetomidine infusion will be administered for intraoperative analgesia Group 2: Remifentanil infusion will be administered for intraoperative analgesia Routine anesthesia protocol in our clinic: patient is induced with fentanyl 1μg/kg IV and propofol 1.5 to 2 mg/kg IV, rocuronium 0.6 mg/kg IV. After putting the patients to sleep, ESP block is applied to the patients for postoperative pain management.

The peroperative analgesia plan will be applied the same to all patients. In this protocol, intravenous paracetamol was determined as 1 g and tramadol was determined as 1 mg/kg. Then it is paracetamol every eight hours and tramadol from PCA.

At the end of the operation, patients' pain levels will be determined and recorded with the Numeric Rating Scale (NRS) system at 4-hour intervals in the first 24 hours postoperatively.

Demographic data to be obtained will include height (cm), weight (kg), age (years), gender, physical condition (ASA) and specific procedure type will be recorded. Patients will be asked about tobacco, alcohol use and drug use. They will also be asked about their medical history, including lung disease, kidney disease, diabetes mellitus, neurological disease, chronic pain conditions, previous surgery or stent placement, and medications. Current preoperative laboratory tests and medication list will be recorded. Preoperative pain scores, NRS, and opioid use will be recorded. Pain levels will be determined and recorded using the Numeric Rating Scale (NRS) system during the first 24 hours postoperatively. Additionally, opioid consumption will be evaluated from the PCA device used postoperatively. Patients excluded for any reason, including technical considerations or contraindications, will be enrolled.

How much intraoperative bleeding occurred, how much blood and blood products were transfused to the patient, and the duration of surgery will be recorded.

F. DATA ANALYSIS Statistical analyzes will be performed using SPSS. Before statistical testing, each continuous variable will be analyzed using the Kolmogorov-Smirnov test to determine whether it has a normal distribution. Continuous data are described as mean (SD) or median (25% and 75% percentiles) and will be analyzed by independent t test or Mann-Whitney U test, respectively. Categorical data were described as frequency or percentage and will be analyzed using the chi-square test. One-way ANOVA with multiple comparison test will be used for comparison between groups. For periods between first PCA triggers, data will be analyzed using the Kaplan-Meier survival method and compare groups using the log-rank test. Results will be expressed as mean ± SD or absolute number, and a P value < 0.05 will be considered statistically significant.

G. NUMBER OF SAMPLES Shobana Rajan et al. Based on their study, investigators calculated a sample size of 37 patients per group by setting alfa equal to 0.005 and beta equal to 0.8.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* 18-75 years old
* ASA Physical Status 1-3;
* Patients planned for lumbar disc surgery

Exclusion Criteria:

* Rejection during registration
* Request for dismissal from employment
* Inability to give informed consent
* Emergency surgery
* Bleeding diathesis
* Chronic use of opioids
* Psychiatric disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | 24 hours
  Patients' opioid consumption on the PCA device will be recorded at 0, 3, 6, 12, 18, and 24 hours postoperatively.

SECONDARY OUTCOMES:
The Numeric Rating Scale (NRS) | 24 hours
  Preoperative period and Postoperative 30th minute, 1st, 6th, 12th, 18th. And at the 24th hour, patients' pain levels and NRS scores will be recorded. At the end of the operation, patients' pain levels will be determined and recorded using the Numeric Rating Scale (NRS) system at intervals in the first 24 hours postoperatively. NRS; It is a pain intensity determination system based on the system of having the person say a point between 0 (no pain), 10 (unbearable pain) and 10 (unbearable pain) to describe his/her pain.

CONTACTS AND LOCATIONS:
Overall Officials: ferdi gülasştı, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Ferdi Gülaştı, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided